CLINICAL TRIAL: NCT05465083
Title: Feasibility of Transvenous Phrenic Nerve Stimulation for Diaphragm Protection in Acute Respiratory Failure: the STIMULUS I Clinical Trial
Brief Title: Feasibility of Transvenous Phrenic Nerve Stimulation for Diaphragm Protection in Acute Respiratory Failure
Acronym: STIMULUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Lungpacer Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-5815; 21-5516 (Other: UHN CAPCR Related ID)
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2023-06

CONDITIONS: Acute Hypoxemic Respiratory Failure; Diaphragm Injury; Lung Injury
MeSH Terms: conditions — Respiratory Insufficiency; Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lungpacer AeroPace Protect System (Experimental): The PNS device used for this study will be the most recent AeroPace central venous catheter from Lungpacer Medical Inc (Vancouver, BC). It is an 8.5F 23cm triple lumen central venous catheter with 30 electrodes arranged in two arrays (distal 9 electrodes intended to capture the right phrenic nerve and the 21 proximal to capture the left phrenic nerve). It is inserted via the left internal jugular or left subclavian vein where it is placed in the proximal superior vena cava (SVC) at or above the cavo-atrial junction.
  The AeroPace system monitors airway pressure to detect ventilator-triggered controlled mechanical breaths and patient-triggered assisted mechanical breaths. In response to detection of native respiratory efforts the PNS lies quiescent.
  Interventions: Device: Lungpacer AeroPace Protect System

INTERVENTIONS:
Device: Lungpacer AeroPace Protect System — AeroPace Catheter will be placed percutaneously into the left internal jugular vein or left subclavian vein and stimulating electrodes mapped for therapy.

SUMMARY:
This is a single-center proof-of-concept clinical trial designed to establish the feasibility of transvenous phrenic-nerve stimulation (PNS) to maintain diaphragm activation over the first 24 hours and for up to seven days of mechanical ventilation in patients who are likely to require more than 48 hours of invasive mechanical ventilation.

DETAILED DESCRIPTION:
The diaphragm is the main muscle of breathing and for most of us therefore is continuously being used (and hence exercised) when in health. When people are unwell with severe breathing difficulties to the degree that their lungs are needing a lot of support from a breathing machine (ventilator) in the intensive care unit (ICU), or are recovering from major lung/chest surgery on a ventilator in ICU, the diaphragm can quickly start to weaken from its inactivity. This means that even when starting to recover from the underlying medical problem, or from the surgery itself, the diaphragm may be unable perform well enough to take over the work of breathing once again. This can lead to not only longer times on the ventilator (time to gradually rebuild diaphragm strength by rehabilitation and physiotherapy) but also therefore longer times in ICU and in hospital with the risk of complications that can be associated with this.

Stimulating the diaphragm by use of a pacemaker (electrical stimulation) is an established treatment for a number of patients with certain types of long-term breathing problems. These pacemakers are permanent and are inserted by invasive surgical methods. More recently however, there have also been a number of studies looking to see if it is possible to safely, temporarily and less invasively stimulate the diaphragm of patients who only have temporary diaphragm inactivity. This has been done either during surgery or during their intensive care stay. A number of methods of temporarily stimulating the diaphragm have been looked at, but the simplest has been to integrate the function of stimulating the nerves (that ultimately control the diaphragm) with a catheter that is frequently placed into a vein in the neck to enable delivery of medications during surgery and in ICU.

ELIGIBILITY:
Group 1: Acute hypoxemic respiratory failure (AHRF)

Inclusion Criteria:

* Age ≥18 years old, and,
* Invasive mechanical ventilation for ≤ 7 days, and,
* Have hypoxemia as defined by one of:
* A PaO2:FiO2 ratio < 300 and PEEP ≥ 5 cm H2O, or
* SpO2:FiO2 < 315% on PEEP ≥ 5 cm H2O in absence of an available arterial blood gas, and in the presence of a reliable Sp)2 trace and a SpO2 < 97%, or
* Are receiving inhaled nitric oxide for acute hypoxemia, or
* Require extracorporeal membrane oxygenation, and,
* Are on controlled mechanical ventilation with no patient-triggered ventilator-delivered breaths with no imminent plan to transition to assisted ventilation within 6 hours, and,
* Are not expected to be liberated from mechanical ventilation within the next 48 hours (from time of enrollment)

Group 2: Pulmonary endarterectomy

Inclusion Criteria:

* Age 18 to 65 years old
* Are listed for pulmonary thromboendarterectomy
* Have pulmonary vascular resistance < 1000 dynes.sec.cm-5

Group 3: Lung transplant

Inclusion Criteria:

* Age 18 years or older
* Are listed for bilateral lung transplant for a primary indication of idiopathic pulmonary fibrosis with no plan for concomitant transplant of other solid organs

All groups

Exclusion Criteria:

* Pregnant or lactating
* Previously diagnosed neuromuscular disorder or known phrenic nerve injury
* BMI >70kg/m2
* Implanted electronic cardiac or neurostimulation device in situ
* Contraindications to left internal jugular or subclavian vein catheterization (e.g., infection over the site, known central venous stenosis, septic thrombophlebitis, left internal jugular ECMO cannula in situ) and/or subclavian vein catheterization (to include poor target vessel)
* Contraindications to esophageal balloon or EMG catheter placement (e.g. active bleeding or high-grade esophageal varices with recent bleeding or banding in previous 14 days, recent esophageal surgery or esophageal rupture)
* Patient transitioning fully to palliative care
* Treating clinician deem enrollment not clinically appropriate for other reason
* Currently being treated in another clinical trial studying an experimental treatment that could affect the study primary outcome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-04 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of placing AeroPace Catheter | 30 days
  Feasibility will be defined as the device being successfully deployed in at least 11 of the 20 patients. Successful deployment of the device defined as:
  * AeroPace Catheter insertion and placement successfully confirmed
  * Initial Catheter electrode mapping/calibration successfully completed
  * Adequate diaphragm activation achieved, defined as hourly Edi level sufficient to generate a Pocc of ≤ -5 cm H2O, for at least 50% of LAPS-PNS stimulated breaths over the first 24 hours after commencing stimulation.
Safety of AeroPace Catheter | 30 days
  The technique will be considered safe if there are no unexpected serious adverse events (USADEs) and the incidence of device- or procedure-related SAEs is below that established in literature.

SECONDARY OUTCOMES:
LAPS-PNS successfully achieved at the time of the mapping/calibration procedure on each of the subsequent days up to the end of the study intervention period | 7 days
The proportion of time that adequate diaphragm activation is maintained during phrenic nerve stimulation and during the absence of phrenic nerve stimulation. | 7 days
  This is defined as the percentage of hours the patient has an Edi ≥ minimum Edi required to maintain Pocc ≤ -5 cm H2O.
The proportion of hours in which the maintenance of diaphragm activation is due to LAPS-PNS rather than endogenous patient respiratory effort. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morris IS, Bassi T, Bellissimo CA, Bootjeamjai P, Roman-Sarita G, de Perrot M, Donahoe L, McRae K, Dianti J, Del Sorbo L, Keshavjee S, Cypel M, Reynolds SC, Dres M, Thakkar V, Mehta N, Brochard L, Ferguson ND, Goligher EC. Continuous On-Demand Diaphragm Neurostimulation to Prevent Diaphragm Inactivity During Mechanical Ventilation: A Phase 1 Clinical Trial (STIMULUS). Am J Respir Crit Care Med. 2025 Aug;211(8):1442-1451. doi: 10.1164/rccm.202407-1483OC. PMID 40043207